CLINICAL TRIAL: NCT02955407
Title: Genetic Predisposition for Reduced Back Muscle Strength and Back Muscle Endurance in Patients With Chronic Non-specific Low Back Pain
Brief Title: Genetic Predisposition for Chronic Non-specific Low Back Pain
Acronym: Backgene
Status: Completed | Type: Observational
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-00647
Record Dates: First submitted 2016-10-06; First posted 2016-11-04 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Low back pain patients: Low back pain since more than 3 months Age: 18-65 Caucasian race
  Interventions: Other: no intervention
- Controls without low back pain: no low back ain Age: 18-65 Caucasian race
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — observational case-control study

SUMMARY:
Patients with inflammatory back pain were shown to differ from healthy controls in genotype of the Angiotensin-converting enzyme (ACE), which regulates vasoconstriction/-dilatation. The aim of this study is to investigate whether genetic reduction of muscle perfusion might be a pathophysiological pathway of how genes influence chronic non-specific low back pain (LBP).

DETAILED DESCRIPTION:
The following genes will be investigated:

* Insertions-/deletions-polymorphism of the angiotensin-converting enzyme (ACE-I/D gene polymorphism; 3 genotypes: ACE-II, ACE-ID, ACE-DD).
* Anti-adhesive extracellular matrix protein Tenascin-C: gene polymorphism rs2104772

The goals of this study are to investigate whether these genotypes correlate with 1) endurance of back muscles, 2) comorbidities such as asthma and diabetes and 3) the risk for LBP as assessed by a LBP-classification tool.

ELIGIBILITY:
Inclusion Criteria:

* 18-65

Exclusion Criteria:

* Spinal surgery
* Spinal fracture
* Inflammation
* Tumour
* Severe chronic disease which make intensive physical activity impossible (osteoporosis, cardiovascular heart diseases)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic low back pain and healthy controls without low back pain.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-09; Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Polymorphism ACE Gene | baseline
Polymorphism Tenascin Gene | baseline

SECONDARY OUTCOMES:
Back muscle endurance in Sorensen test | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Martin Flück, Professor, Study Director — Balgrist University Hospital
Locations (1):
- Balgrist University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vaughan D, Huber-Abel FA, Graber F, Hoppeler H, Fluck M. The angiotensin converting enzyme insertion/deletion polymorphism alters the response of muscle energy supply lines to exercise. Eur J Appl Physiol. 2013 Jul;113(7):1719-29. doi: 10.1007/s00421-012-2583-6. Epub 2013 Feb 9. PMID 23397151
- [Background] Shehab DK, Al-Jarallah KF, Al-Awadhi AM, Al-Herz A, Nahar I, Haider MZ. Association of angiotensin-converting enzyme (ACE) gene insertion-deletion polymorphism with spondylarthropathies. J Biomed Sci. 2008 Jan;15(1):61-7. doi: 10.1007/s11373-007-9203-1. Epub 2007 Aug 23. PMID 17713861